CLINICAL TRIAL: NCT02422160
Title: Vision Outcomes Using Quantitative Optical Coherence Tomography Evaluation in Age Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theodore Leng, Principle Investigator, Stanford University
Other Study IDs: 33624
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions are planned — No interventions are planned

SUMMARY:
The investigators have developed an image analysis method that can predict the likelihood that a patient with age related macular degeneration (AMD) will progress within 1 year, based on computerized analysis of optical coherence tomography (OCT) images that are routinely acquired in clinical practice on each patient visit to the ophthalmologist. The investigators' goal is to evaluate whether this method will improve the ability to detect AMD earlier and improve visual outcomes in AMD patients by assigning patient risk categories and having patients come back for follow up based on those categories.

ELIGIBILITY:
Inclusion Criteria:

* Non-exudative age-related macular degeneration

Exclusion Criteria:

* Exudative age-related macular degeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-exudative age-related macular degneration
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | Two Years

CONTACTS AND LOCATIONS:
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States